CLINICAL TRIAL: NCT01374555
Title: Validation of the CardioSond Sonospectrographic Digital Electronic Stethoscope in Diagnosing Coronary Artery Disease Versus CT Angiography
Brief Title: Evaluation of the CardioSond Electronic Stethoscope in the Detection of Coronary Artery Disease
Status: Terminated | Type: Observational
Why Stopped: Inconsistent data taken from Phase I cohort
Sponsor: SonoMedica, Inc. (Industry)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: SM-C103; 2010-153 (Other: Medstar Research Institute)
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2013-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed to evaluate the predictive accuracy of the CardioSond digital electronic stethoscope in the detection of coronary artery disease (CAD) in patients with and without known disease who are referred to cardiac computed tomography angiography (CT scans).

DETAILED DESCRIPTION:
The CardioSond is a noninvasive medical device which detects heart sounds using ultrasensitive acoustic technology. The CardioSond produces a flow micro bruit score which is used to determine the likelihood of coronary artery disease.

The CardioSond exam will be given to patients two times: once prior to administration of vasodilators and potential beta blockade agents as part of the normal cardiac CT angiography protocol and again immediately post CT angiography. No other data will be taken on the patient and the patients involvement in the study will cease after data collection.

CT angiography data will be analyzed at a core lab at Medstar Research Institute and withheld from SonoMedica until all CardioSond acoustic data is analyzed and flow micro bruit scores are determined.

A data review panel lead by the principal investigator will examine the results of both the CardioSond and CT angiography data to determine the comparative accuracy of the CardioSond in detecting CAD in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent.

Exclusion Criteria:

* Inability to provide informed consent
* History of prior myocardial infarction, percutaneous coronary intervention (i.e. stents) or coronary artery bypass graft surgery
* Heart rate over 70 beats per minute post beta blockade
* Artery calcification resulting in non-diagnostic CT angiographic images
* Supraventricular or ventricular arrhythmias that would be expected to affect CT angiography image quality (e.g. atrial fibrillation, atrial flutter, ventricular tachycardia, bigeminy and trigeminy). Patients with isolated premature atrial contraction and premature ventricular contractions may enroll
* Any pulmonary condition that would create abnormal physical findings that would interfere with the fidelity of the cardiac sound recordings (e.g. obstructive pulmonary disease, such as asthma or COPD, with audible wheezing)
* Presence of audible aortic or pulmonic diastolic murmurs, tricuspid or mitral flow diastolic murmurs or continuous murmurs
* Any chest wall configuration preventing adequate contact between the CardioSond acoustic recording sensor and precordium
* Any medical condition that would be expected to affect CT angiography image quality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be sourced from patients presenting for cardiac CT angiography who meet inclusion / exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2010-09-29 (Actual); Primary Completion 2011-04-27 (Actual); Study Completion 2011-04-27 (Actual)

PRIMARY OUTCOMES:
Determine the comparative diagnostic accuracy of the CardioSond digital electronic stethoscope versus CT angiography in detecting CAD, as defined as a stenosis of a major epicardial coronary artery of 50% or greater. | Patient participation will be limited to the day of their CT angiography exam (day 1). Patients will receive two seperate CardioSond examinations which on average takes approximately 20 minutes.
  The CardioSond digital electronic stethoscope's flow micro bruit score will be used as an indication of probability of disease in patients with and without known disease and compared to the results of CT angiography.

SECONDARY OUTCOMES:
Determine the effects of vasodilators and beta blockade on CardioSond digital electronic stethoscope data results on data taken post CT angiography. | Patient participation will be limited to the day of their CT angiography exam (day 1). Patients will receive two seperate CardioSond examinations which on averages takes approximately 20 minutes.
  The patient's flow micro bruit scores from each CardioSond examination (one pre CT angiography and one post CT angiography) will be compared to each other to assess the effects on the score of vasodilators administered as part of the CT angiography exam.

CONTACTS AND LOCATIONS:
Overall Officials: Allen J. Taylor, M.D., Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States